CLINICAL TRIAL: NCT02292797
Title: Assessment of the Prevalence of Rosacea in the General Population
Brief Title: Assessment of the Rosacea Prevalence in the General Population
Acronym: RISE
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: RD.03.SPR.29104
Record Dates: First submitted 2014-10-14; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prevalence assessment — Assessment of the prevalence of rosacea in the general population per country using subject questionnaire and dermatologist diagnosis

SUMMARY:
Multi-centre interventional cross-sectional prevalence study Assessment of the Rosacea Prevalence in the General Population.

DETAILED DESCRIPTION:
Primary objective:

Assessment of the prevalence of rosacea in the general population per country using subject questionnaire and dermatologist diagnosis

ELIGIBILITY:
Part I

Inclusion Criteria:

The following subjects will be included in the study:

* Subjects aged 18 to 65 years old from the general population
* Subjects who are willing to complete the questionnaires

Part II

Inclusion Criteria:

The following subjects will be included in Part II of the study:

* Subjects who screened positive for rosacea during the first part of the study and selected by random method
* Subjects who gave their informed consent to participate in Part II of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part I:
  Subjects will be screened from the general population by questionnaires mainly focusing on detection of signs and symptoms of rosacea.
  Subjects' answers will be submitted to a pre-defined algorithm to identify the potential subjects with rosacea (screened positive for rosacea, Screened R+).
  Part II:
  A subgroup of subjects (100 maximum per country) will be randomly selected among those who screened positive for rosacea and will be referred to the closest investigational site (dermatologist practice).
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
percentage of subjects with rosacea diagnosis confirmed | general population will be surveyed over an expected average duration of 6 months
  estimation of the percentage of rosacea patients in the general population

CONTACTS AND LOCATIONS:
Overall Officials: Fabien AUDIBERT, Bsc, Study Director — Galderma R&D